CLINICAL TRIAL: NCT05647980
Title: Transmural Collaborative Care Model for Cardiovascular Risk Management (CVRM) and Medication Review for Patients Using Antipsychotics: a Cluster Randomised Stepped Wedge Trial
Brief Title: Transmural Collaborative Care Model for CVRM and Medication Review for Patients Using Antipsychotics
Acronym: TACTIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Onze Huisartsen BV. (Unknown)
Responsible Party: Principal Investigator, E. Bischoff, Principle investigator, Radboud University Medical Center
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10140021910502
Record Dates: First submitted 2022-09-20; First posted 2022-12-13 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Mental Disorders, Severe
Keywords: Primary health care; Antipsychotics; Cardiovascular risk; Collaborative care; Deprescribing; Off label
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Incomplete stepped wedge cluster randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACTIC (Experimental): Participants in the TACTIC intervention will be provided a 3-step approach, i.e.
  1. an online information video to inform patients about the cardiovascular risks of antipsychotic use and the procedures of the multidisciplinary meeting
  2. a multidisciplinary meeting with their general practitioner, the primary care nurse, a psychiatrist, and an experience expert to discuss cardiovascular risk and side effect and to provide personalised treatment options
  3. a consultation with their general practitioner to translate treatment options into an individualised treatment plan including lifestyle and medication treatment and monitoring frequency, based on shared-decision making
  Interventions: Other: TACTIC
- Care as usual (No Intervention): Care as usual, i.e. renewal of prescriptions for antipsychotics by the general practitioner without multidisciplinary treatment advice and without the use of scheduled and structured monitoring visits.

INTERVENTIONS:
Other: TACTIC — Participants execute the three steps of TACTIC Participants fill in questionnaires Participants take laboratory and biometric tests to measure their cardiovascular risk
  Arms: TACTIC

SUMMARY:
Currently, monitoring of usage and effects of antipsychotic treatment and cardiovascular risk screening in patients with severe mental illness or antipsychotic treatment is not sufficient.

A transmural collaborative care model for cardiovascular risk management and medication review for patients using atypical antipsychotics in general practice (TACTIC) was developed. This trial aims to assess the effectiveness of TACTIC regarding predicted cardiovascular risk and mental quality of life.

DETAILED DESCRIPTION:
It is well established that patients with severe mental illness and patients treated with atypical antipsychotics have excess metabolic dysfunction and are at an increased risk of cardiovascular disease. Currently, monitoring of usage and effects of antipsychotic treatment and cardiovascular risk screening in patients with severe mental illness or antipsychotic treatment is not sufficient. General practitioners experience barriers regarding knowledge, collaboration with psychiatrists, and patient compliance. To overcome these barriers a transmural collaborative care model for cardiovascular risk management and medication review for patients using atypical antipsychotics in general practice (TACTIC) was developed. TACTIC is a one-time transmural intervention comprising three steps: 1) an online information video to inform patients about the cardiovascular risks of antipsychotic use and the procedures of the multidisciplinary meeting, 2) a multidisciplinary meeting with the patient to review his or her antipsychotic use and cardiovascular risk and to provide tailored treatment advice, and 3) a follow-up contact with the general practitioner to translate the treatment advice into an individualised action plan through shared decision making.

This trial aims to assess the effectiveness of TACTIC regarding predicted cardiovascular risk and mental quality of life.

ELIGIBILITY:
Inclusion Criteria:

* using atypical antipsychotic medication for at least 3 months at baseline
* the atypical antipsychotic medication is prescribed by the general practitioner
* a 10-year cardiovascular risk of at least 5% (as measured with QRISK3 score) at baseline

Exclusion Criteria:

* diagnosis of dementia or organic psychosis
* diagnosis of cardiovascular disease (acute myocardial infarction, acute coronary syndrome, heart failure, ischemic stroke, transient ischemic attack, peripheral artery disease, aortic aneurysm or a revascularization procedure, i.e. percutaneous coronary intervention or coronary artery bypass grafting)

Ages: 25 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The change in QRISK3 score as measured with the QRISK3 calculator (https://qrisk.org/three/) | Measurements at baseline, at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  The risk score of developing cardiovascular disease over the next 10 years is estimated using the QRISK®3 algorithm (https://qrisk.org/three/), which calculates a person's ten-year risk of cardiovascular disease by taking multiple risk parameters into account. A higher score means a higher risk. Risks may vary between 0% and 100%. The parameter Townsend deprivation score will be set to 0 (as advised by its developers), meaning neither deprived nor affluent, as this score does not apply to the Dutch population.
The change in Mental Health, as measured with the Mental Health Inventory questionnaire | Measurements at baseline, at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  Mental Health is measured using the five-item version of the Mental Health Inventory (MHI) questionnaire. The MHI-5 is a derivative of the 36-item short form (SF-36) health survey, and assesses symptoms of depression and anxiety, loss of behavioural or emotional control, and psychological well-being in the prior four weeks. Scores range from 0 to 100, lower scores are worse, and patients with a score ≥60 are considered mentally healthy.

SECONDARY OUTCOMES:
The change in Quality of Life (QoL) as measured with the EuroQuality of Life Five Dimensions (EQ-5D-5L) questionnaire | Measurements at baseline, at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  QoL is measured using the EuroQuality of Life Five Dimensions (EQ-5D-5L) questionnaire, which measures generic quality of life on 5 domains with a 5-point Likert scale. A higher score means a worse healt state in each domain, with a maximum of 5 points.
The change in Side effects of antipsychotic medication, as measured with the Liverpool University Neuroleptic Side Effect Rating Scale (LUNSERS) questionnaire | Measurements at baseline, at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  The side effects of antipsychotic medication is measured using the Liverpool University Neuroleptic Side Effect Rating Scale (LUNSERS) questionnaire, which assesses side effects of neuroleptic drugs. It has been designed to enable the client to make the rating themselves but can also be administered by mental health workers if the client is unable to complete it. The scale consists of 41 known side effects of neuroleptics. Each 'side-effect' listed is scored on a five point rating scale of 0 - 4, i.e. 0 = 'Not at all' and 4 = Very much. A higher total score means more side-effects. Maximum total score is 84
The change in Client Satisfaction, as measured with the 8-item Client Satisfaction Questionnaire (CSQ-8) | At 5 months from baseline
  Client Satisfaction with care is measured using the CSQ-8, an 8-item questionnaire using a 4-point Likert scale. The sum of 8 sub-scores about different aspects of received care can vary between 8 and 32. Higher scores mean higher satisfaction.
The change in risk score of developing cardiovascular disease over the next 10 years including a Dutch deprivation score | Measurements at baseline, at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  The risk estimation of the QRISK3 score is based on several parameters including the Townsend deprivation score. For the primary outcome the score will be set to 0, as the original score does not apply to the Dutch population. For this secondary outcome the QRISK3 score will be calculated including a Dutch deprivation index. A higher score means a higher risk. Risks may vary between 0% and 100%.
The change in QRISK3 score as proportion of the maximum achievable change in QRISK3 score | Measurements at baseline baseline at 5, 10, 15 and 20 months (depending on the specific wave in the stepped-wedge trial in which follow-up starts)
  The change in QRISK3 score as a proportion of the maximum achievable change in QRISK3 score is the change in QRISK3 score that has been achieved at the end of follow-up divided by the change in QRISK3 score that could have been achieved when all modifiable risk factors would have been improved. The proportional score may be 1.0 (actual change equals maximum achievable change) or less.
The change in costs related to health care | 1-20 months (depending on the duration of follow-up which differs between the waves in the stepped-wedge trial.
  Costs include health care utilization, such as medication use, visits to the general practice, visits to relevant medical specialists, hospitalisation. Costs will be calculated during follow-up time and will be compared with the same period of time prior to start of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Erik E Bischoff, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical centre, Dept. Primary and Community Care, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The Research Information Services (RIS) interface, specifically developed for the Radboud University Nijmegen, will also be used to register and archive our data in the certified DANS EASY archive of KNAW and NWO.
Supporting Information: Study Protocol, SAP
Time Frame: 1-March-2023 until 1-March 2037
Access Criteria: Data are available on request of the principle investigator

REFERENCES:
- [Background] Bischoff EWMA, Jakobs KM, Assendelft WJJ. Cardiovascular risk management in patients using antipsychotics: it is time to take action. BMC Med. 2020 Nov 2;18(1):339. doi: 10.1186/s12916-020-01811-7. No abstract available. PMID 33131496
- [Background] Jakobs KM, Posthuma A, de Grauw WJC, Schalk BWM, Akkermans RP, Lucassen P, Schermer T, Assendelft WJJ, Biermans MJC. Cardiovascular risk screening of patients with serious mental illness or use of antipsychotics in family practice. BMC Fam Pract. 2020 Jul 29;21(1):153. doi: 10.1186/s12875-020-01225-7. PMID 32727372
- [Background] Jakobs K, Lautan L, Lucassen P, Janzing J, van Lieshout J, Biermans MCJ, Bischoff EWMA. Cardiovascular risk management in patients with severe mental illness or taking antipsychotics: A qualitative study on barriers and facilitators among dutch general practitioners. Eur J Gen Pract. 2022 Dec;28(1):191-199. doi: 10.1080/13814788.2022.2092093. PMID 35796600
- [Derived] Jakobs KM, van den Brule-Barnhoorn KJ, van Lieshout J, Janzing JGE, Cahn W, Kievit W, Teerenstra S, van den Muijsenbergh M, Biermans MCJ, Bischoff EWMA. Transmural collaborative care model for cardiovascular risk management and medication review in patients using antipsychotics in primary care (TACTIC): A study protocol of an incomplete stepped wedge cluster randomized trial. Contemp Clin Trials Commun. 2025 Jan 9;44:101418. doi: 10.1016/j.conctc.2024.101418. eCollection 2025 Apr. PMID 39897941

DOCUMENTS (1):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT05647980/Prot_000.pdf